CLINICAL TRIAL: NCT00603538
Title: Phase 1, Dose Escalation Study of CP-751,871 in Combination With Carboplatin and Paclitaxel in Previously Untreated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Study of CP-751,871 in Combination With Carboplatin and Paclitaxel in Advanced Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021019; Japan CTPN 19-2409
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: CP-751,871, Non-small cell lung cancer, Phase 1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — figitumumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CP-751,871 (Experimental)
  Interventions: Drug: CP-751,871 + carboplatin + paclitaxel

INTERVENTIONS:
Drug: CP-751,871 + carboplatin + paclitaxel — Chemotherapy (carboplatin and paclitaxel) and CP-751,871 (6, 10 or 20mg/kg) will be administered by intravenous infusion every three weeks.

SUMMARY:
Investigate safety, tolerability and pharmacokinetics of CP-751,871 when given in combination with carboplatin and paclitaxel in patients with advanced non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced non-small cell lung cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Any prior treatment for non-small cell lung cancer
* Brain metastases
* With diabetes

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Derived] Goto Y, Sekine I, Tanioka M, Shibata T, Tanai C, Asahina H, Nokihara H, Yamamoto N, Kunitoh H, Ohe Y, Kikkawa H, Ohki E, Tamura T. Figitumumab combined with carboplatin and paclitaxel in treatment-naive Japanese patients with advanced non-small cell lung cancer. Invest New Drugs. 2012 Aug;30(4):1548-56. doi: 10.1007/s10637-011-9715-4. Epub 2011 Jul 13. PMID 21748299
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021019&StudyName=Study%20of%20CP-751%2C871%20in%20Combination%20with%20Carboplatin%20and%20Paclitaxel%20in%20Advanced%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-751,871 6 mg/kg in Combination With Chemotherapy Agents: CP-751,871 6 mg/kg was administered intravenously on Day 1 of each 21-day cycle in combination with following chemotherapy; paclitaxel 200 mg/m^2 was administered intravenously over 3 hours, then carboplatin AUC 6 was administered intravenously over 30 minutes or longer prior to the CP-751,871 infusion. Study treatment was repeated up to 4 cycles, unless disease progression or unacceptable toxicity was observed, and then up to 6 cycles if the participant showed response or stable disease at the end of Cycle 4 and agreed on additional treatment.
- CP-751,871 10 mg/kg in Combination With Chemotherapy Agents: CP-751,871 10 mg/kg was administered intravenously on Day 1 of each 21-day cycle in combination with following chemotherapy; paclitaxel 200 mg/m^2 was administered intravenously over 3 hours, then carboplatin AUC 6 was administered intravenously over 30 minutes or longer prior to the CP-751,871 infusion. Study treatment was repeated up to 4 cycles, unless disease progression or unacceptable toxicity was observed, and then up to 6 cycles if the participant showed response or stable disease at the end of Cycle 4 and agreed on additional treatment.
- CP-751,871 20 mg/kg in Combination With Chemotherapy Agents: CP-751,871 20 mg/kg was administered intravenously on Day 1 of each 21-day cycle in combination with following chemotherapy; paclitaxel 200 mg/m^2 was administered intravenously over 3 hours, then carboplatin AUC 6 was administered intravenously over 30 minutes or longer prior to the CP-751,871 infusion. Study treatment was repeated up to 4 cycles, unless disease progression or unacceptable toxicity was observed, and then up to 6 cycles if the participant showed response or stable disease at the end of Cycle 4 and agreed on additional treatment.
Period: Overall Study
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Started | 6 | 7 (Including one participant who discontinued from the study prior to CP-751,871 administration.) | 6
Completed | 3 | 3 | 4
Not Completed | 3 | 4 | 2
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Objective progression or relapse | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents | Total
Number analyzed (Participants) | 6 | 7 | 6 | 19
Age, Customized [Number; unit: participants]
  20 to 44 years | 0 | 5 | 1 | 6
  45 to 64 years | 4 | 2 | 2 | 8
  >=65 years | 2 | 0 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 7
  Male | 3 | 4 | 5 | 12
ECOG Performance Status [Number; unit: participants] — ECOG = Eastern Cooperative Oncology Group. ECOG Grade: 0: Fully active. 1: Ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of all selfcare. 3: Capable of limited selfcare, confined to bed or chair more than 50% of waking hours. 4: Completely disabled, no selfcare, totally confined to bed or chair. 5: Dead.
  participants
    Score 0 | 5 | 7 | 4 | 16
    Score 1 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: A DLT was defined as any one of the following adverse events observed in Cycle 1 which was considered as related to CP-751,871 combination therapy; 1) >=Grade 3 gastrointestinal toxicity, hyperglycemia and/or fatigue despite the use of adequate/optimal medical intervention, 2) Any other >=Grade 3 toxicity not classified under CTCAE blood/bone marrow, or 3) Grade 4 neutropenia that persisted for >=7 consecutive days or was complicated by fever (defined as a body temperature >38.0 Celsius degree), 4) Grade 3 thrombocytopenia which needed blood transfusion or Grade 4 thrombocytopenia.
Time Frame: Cycle 1
Population: DLT Evaluation Set comprised of participants who were treated with CP-751,871. One participant in the 10 mg/kg cohort who discontinued from the study due to an adverse event occurred prior to CP-751,871 administration was excluded from this analysis set.
Measure: Number; unit: participants
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 6 | 6 | 6
participants | 1 | 2 | 0

2. Secondary Outcome: Maximum Observed Concentration (Cmax) of CP-751,871
Time Frame: Cycles 1 and 4 at prior to dosing of CP-751,871 (Day 1), and 1, 24, 72 and 168 (Day 8) hours after end of CP-751,871 infusion
Population: The Pharmacokinetics Analysis Set was defined as all participants who started treatment and had sufficient information for estimation of pharmacokinetic parameters.
  n = the number of participants analyzed
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 6 | 6 | 6
mg/L
  Cycle 1 (n=6,6,6) | 113 (16) | 197 (33) | 485 (59)
  Cycle 4 (n=4,4,5) | 178 (35) | 294 (61) | 550 (89)

3. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Cycle 1 : prior to CP-751,871 (Day 1) dosing, and 1, 24, 72 and 168 (Day 8) hours after end of CP-751,871 infusion
Population: Participants with sufficient sampling to capture the terminal disposition phase were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 4 | 1 | 4
hours | 264 (38.9) | NA (NA) — Mean was not calculated because there was only 1 participant to be analyzed. | 248 (30.1)

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Day 22 (AUC0-day22)
Description: AUC(0-day22) : AUC from time zero (Day 1) to Day 22, where Day 22 is the nominal time (504 hours) of the predose sampling for the next cycle. AUC(0-day22) was calculated using the linear/log trapezoidal method.
Time Frame: Cycle 1: prior CP-751,871 (Day 1) to dosing, and 1, 24, 72 and 168 (Day 8) hours after end of CP-751,871 infusion
Population: The Pharmacokinetics Analysis Set was defined as all participants who started treatment and had sufficient information for estimation of pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 6 | 6 | 6
mg*h/L | 22400 (4050) | 36700 (10400) | 82700 (11200)

5. Secondary Outcome: Area Under the Plasma Concentration Curve From Time Zero to Tau (AUCtau)
Description: AUCtau: AUC from time zero to tau, the dosing interval, where tau is the actual time of the predose sampling for the next cycle. AUCtau was calculated using the linear/log trapezoidal method.
Time Frame: Cycle 4: prior to CP-751,871 (Day 1) dosing , and 1, 24, 72 and 168 (Day 8) hours after end of CP-751,871 infusion
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg*h/mL
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 2 | 2 | 2
mg*h/mL | NA (NA) — Mean was not calculated because there were only 2 participants who had estimable AUCtau at Cycle 4. | NA (NA) — Mean was not calculated because there were only 2 participants who had estimable AUCtau at Cycle 4. | NA (NA) — Mean was not calculated because there were only 2 participants who had estimable AUCtau at Cycle 4.

6. Secondary Outcome: Observed Accumulation Ratio (Rac)
Description: The ratio of Cycle 4 AUCtau to Cycle 1 AUCtau
Time Frame: Cycle 1 and Cycle 4: prior to CP-751,871 (Day 1) dosing, and 1, 24, 72 and 168 (Day 8) hours after end of CP-751,871 infusion
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 2 | 2 | 2
ratio | NA (NA) — Mean was not calculated because there were only 2 participants who had estimable Rac at Cycle 4. | NA (NA) — Mean was not calculated because there were only 2 participants who had estimable Rac at Cycle 4. | NA (NA) — Mean was not calculated because there were only 2 participants who had estimable Rac at Cycle 4.

7. Secondary Outcome: Serum Concentrations of Total Insulin-like Growth Factor 1 (IGF-1)
Description: IGF-1 is one of the IGF-axis related biomarkers.
Time Frame: Day 1 of Cycles 1 to 6, Day 8 of Cycles 1 to 4, and end of study
Population: Safety Analysis Set was defined as all participants who have received at least one dose of the study medication. n = number of subjects evaluable.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 6 | 7 | 6
ng/L
  Cycle 1 Day 1 (n=6,7,6) | 126.2 (54.0) | 167.7 (64.2) | 136.8 (45.4)
  Cycle 1 Day 8 (n=6,6,6) | 518.3 (199.3) | 611.7 (210.9) | 493.8 (114.6)
  Cycle 2 Day 1 (n=6,5,6) | 579.8 (172.8) | 773.6 (207.1) | 649.5 (104.8)
  Cycle 2 Day 8 (n=6,5,6) | 709.0 (205.4) | 819.8 (214.0) | 544.7 (157.0)
  Cycle 3 Day 1 (n=5,4,6) | 649.8 (129.8) | 864.0 (134.2) | 706.0 (174.3)
  Cycle 3 Day 8 (n=5,4,6) | 774.2 (203.4) | 765.5 (43.6) | 698.0 (97.1)
  Cycle 4 Day 1 (n=4,4,5) | 812.5 (299.5) | 867.3 (224.1) | 634.4 (66.7)
  Cycle 4 Day 8 (n=4,4,5) | 784.5 (148.5) | 904.8 (207.2) | 749.0 (168.5)
  Cycle 5 Day 1 (n=2,2,2) | 908.0 (199.4) | 788.5 (187.4) | 565.0 (97.6)
  Cycle 6 Day 1 (n=2,2,1) | 835.0 (118.8) | 927.0 (2.8) | 695.0 (NA) — Only one participant was available for analysis
  End of treatment (n=5,6,6) | 562.8 (194.5) | 830.3 (304.9) | 655.2 (136.3)

8. Secondary Outcome: Serum Concentrations of Total Insulin-like Growth Factor Binding Protein-3 (IGF-BP-3)
Description: IGF-BP3 is one of the IGF-axis related biomarkers.
Time Frame: Day 1 of Cycles 1-6, Day 8 of Cycles 1-4, and end of treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 6 | 7 | 6
mg/L
  Cycle 1 Day 1 (n=6,7,6) | 2.38 (0.82) | 2.26 (0.59) | 2.55 (0.39)
  Cycle 1 Day 8 (n=6,6,6) | 4.35 (1.41) | 4.20 (0.67) | 3.85 (0.46)
  Cycle 2 Day 1 (n=6,5,6) | 5.12 (1.78) | 5.68 (0.29) | 5.25 (1.93)
  Cycle 2 Day 8 (n=6,5,6) | 6.53 (2.26) | 6.26 (1.18) | 4.63 (0.71)
  Cycle 3 Day 1 (n=5,4,6) | 6.08 (2.23) | 6.78 (1.44) | 5.07 (1.49)
  Cycle 3 Day 8 (n=5,4,6) | 4.66 (1.82) | 5.93 (0.75) | 5.30 (1.04)
  Cycle 4 Day 1 (n=4,4,5) | 5.13 (1.36) | 5.18 (1.04) | 4.32 (0.38)
  Cycle 4 Day 8 (n=4,4,5) | 5.10 (1.55) | 4.95 (2.12) | 4.44 (0.53)
  Cycle 5 Day 1 (n=2,2,2) | 3.45 (1.63) | 5.35 (3.89) | 3.90 (1.27)
  Cycle 6 Day 1 (n=2,2,1) | 5.75 (1.77) | 6.85 (1.20) | 3.20 (NA) — Only one participant was available for analysis
  End of treatment (n=5,6,6) | 4.66 (0.74) | 5.93 (0.75) | 4.63 (0.80)

9. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) Specific to CP-751,871 Following an Intravenous Infusion of CP-751,871.
Description: The screening assay for anti-CP-751,871 antibodies was performed.
Time Frame: Day 1 of Cycles 1 (predose) and 4, and end of study
Population: All participants were screened for the ADA.
Measure: Number; unit: participants
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 6 | 7 | 6
participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Objective Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: Baseline up to 6 cycles (1 cycle = 21 days)
Population: Full Analysis Set (FAS) was defined as all participants who met all of the following criteria; 1) Those who were diagnosed with NSCLC, 2) Those who received at least one dose of the study treatment, and 3) Those who had efficacy data after the start of the study treatment.
Measure: Number; unit: participants
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 6 | 6 | 6
participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 1 | 3 | 3
  Objective Response (CR+PR) | 1 | 3 | 3

11. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is the period from the registration to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Time Frame: Baseline up to 6 cycles (1 cycle = 21 days)
Population: Number of participants with defined event (all causality death or PD) was too few to conduct summary analysis.
Groups:
- CP-751,871 6mg/kg in Combination With Chemotherapy Agents: CP-751,871 6mg/kg was administered intravenously on Day 1 of each 21-day cycle in combination with following chemotherapy agents; paclitaxel 200 mg/m^2 was administered intravenously over 3 hours, then carboplatin AUC 6 was administered intravenously over 30 minutes or longer prior to the CP-751,871 infusion. Study treatment was repeated up to 4 cycles, unless disease progression or unacceptable toxicity was observed, and then up to 6 cycles if the participant showed response or stable disease at the end of Cycle 4 and agreed on additional treatment.
- CP-751,871 10mg/kg in Combination With Chemotherapy Agents: CP-751,871 10mg/kg was administered intravenously on Day 1 of each 21-day cycle in combination with following chemotherapy agents; paclitaxel 200 mg/m^2 was administered intravenously over 3 hours, then carboplatin AUC 6 was administered intravenously over 30 minutes or longer prior to the CP-751,871 infusion. Study treatment was repeated up to 4 cycles, unless disease progression or unacceptable toxicity was observed, and then up to 6 cycles if the participant showed response or stable disease at the end of Cycle 4 and agreed on additional treatment.
- CP-751,871 20mg/kg in Combination With Chemotherapy Agents: CP-751,871 20mg/kg was administered intravenously on Day 1 of each 21-day cycle in combination with following chemotherapy agents; paclitaxel 200 mg/m^2 was administered intravenously over 3 hours, then carboplatin AUC 6 was administered intravenously over 30 minutes or longer prior to the CP-751,871 infusion. Study treatment was repeated up to 4 cycles, unless disease progression or unacceptable toxicity was observed, and then up to 6 cycles if the participant showed response or stable disease at the end of Cycle 4 and agreed on additional treatment.
Arm/Group | CP-751,871 6mg/kg in Combination With Chemotherapy Agents | CP-751,871 10mg/kg in Combination With Chemotherapy Agents | CP-751,871 20mg/kg in Combination With Chemotherapy Agents
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For serious adverse events, up to 150 days after the last administration of the study drugs
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents (N=6) | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents (N=7) | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents (N=6)
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 6 mg/kg in Combination With Chemotherapy Agents (N=6) | CP-751,871 10 mg/kg in Combination With Chemotherapy Agents (N=7) | CP-751,871 20 mg/kg in Combination With Chemotherapy Agents (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 5 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 5 | 4
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 6
Stomatitis (Gastrointestinal disorders) | 4 | 4 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1
Fatigue (General disorders) | 3 | 2 | 4
Feeling hot (General disorders) | 0 | 1 | 0
Hangover (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Gingival infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Trichophytosis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 2 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 3
Blood glucose increased (Investigations) | 2 | 3 | 5
Blood magnesium increased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 2
Blood potassium increased (Investigations) | 2 | 0 | 2
Blood sodium decreased (Investigations) | 2 | 0 | 3
Blood uric acid increased (Investigations) | 1 | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 2 | 3 | 1
Haemoglobin decreased (Investigations) | 5 | 3 | 5
Lymphocyte count decreased (Investigations) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 3 | 1 | 5
Platelet count decreased (Investigations) | 2 | 0 | 5
Weight decreased (Investigations) | 2 | 1 | 4
White blood cell count decreased (Investigations) | 3 | 1 | 5
Anorexia (Metabolism and nutrition disorders) | 3 | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 5 | 6
Insomnia (Psychiatric disorders) | 2 | 3 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 6 | 6
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 5 | 3
Flushing (Vascular disorders) | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.